CLINICAL TRIAL: NCT03553186
Title: Topical Tranexamic Acid as a Adjunct to Intravenous Tranexamic Acid in Adult Spinal Deformity Surgery
Brief Title: Tranexamic Acid in Adult Spinal Deformity Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0920
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Spinal Deformity; Degenerative Lumbar Spinal Stenosis; Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Simple blinded randomization will occur by the pharmacy prior to distribution of the intervention drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ivTXA + topical TXA (Experimental): TXA lavage solution (200 cc sterile normal saline + 5 g tranexamic acid 100mg/ml (50cc)) will be poured into the surgical field and left in contact for five minutes. This will occur after instrumentation. Excess solution will be suctioned away using a non-cell saver suction.
  IV txa will be given as (5mg/ml) loading dose (20mg/kg) over 15 minutes followed by 2 mg/kg/hr maintenance dosing as per hospital protocol
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- IV TXA + topical placebo (Placebo Comparator): Placebo solution (200 cc sterile normal saline + placebo TXA ampule (normal saline) (50cc)) will be poured into the surgical field and left in contact for five minutes. This will occur after pedicle screw instrumentation. Excess solution will be suctioned away using a non-cell saver suction.
  IV txa will be given as (5mg/ml) loading dose (20mg/kg) over 15 minutes followed by 2mg/kg/hr maintenance dosing as per hospital protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — TXA lavage solution (200 cc sterile normal saline + 5 g tranexamic acid 100mg/ml (50cc)) will be poured into the surgical field and left in contact for five minutes. This will occur after instrumentation. Excess solution will be suctioned away using a non-cell saver suction.
  Other Names: Intervention group
  Arms: ivTXA + topical TXA
Drug: Placebo — Placebo solution (200 cc sterile normal saline + placebo TXA ampule (50cc)) will be poured into the surgical field and left in contact for five minutes. This will occur after pedicle screw instrumentation. Excess solution will be suctioned away using a non-cell saver suction.
  Other Names: Control group
  Arms: IV TXA + topical placebo

SUMMARY:
Posterior spinal surgery for adult deformity is associated with high incidence of blood loss and need for blood transfusion and intraoperative blood salvage, with associated increased cost and risk for perioperative complications. Tranexamic acid (TXA) is relatively inexpensive anti-fibrinolytic agent that has been proven effective for decreasing intraoperative blood loss in various surgical specialties. Intravenous TXA (ivTXA) is routinely used at our institution for adult spinal deformity cases. Meanwhile, topical TXA (tTXA) is an attractive alternative/adjunct to ivTXA used with good results in orthopedic arthroplasty and cardiac surgery. To the investigators' knowledge, no data exists in the literature on the use of tTXA in either adult or pediatric spinal deformity surgery. The goal of this study is to determine the role tTXA has an adjunct to ivTXA in decreasing perioperative blood loss, drainage, transfusion requirements and length of stay following adult deformity spine surgery.

DETAILED DESCRIPTION:
Blood loss is a significant issue in spinal deformity surgery, often requiring allogenic blood transfusion and/or intraoperative blood salvage and leading to increased risk of postoperative morbidity, increased length of stay, and higher total hospital costs. Tranexamic acid is an antifibrinolytic agent that is used in many surgical specialties to prevent perioperative blood loss. Intravenous (ivTXA) dosing has proven effective in reducing blood loss and perioperative transfusion in spinal surgery, while the topical (tTXA) form has been shown to be at least non-inferior to IV transfusion in the total arthroplasty literature. Intravenous TXA is routinely used at the investigators' institution in spinal deformity cases, but even with ivTXA infusion, perioperative blood loss remains a significant issue, with total estimated and calculated blood loss between ~1500-3000 mL. Usage of local tTXA in addition to ivTXA may provide additional benefits including an additive effect on decreasing blood loss, allowing for lowered dosages of ivTXA, decreasing risks associated with systemic exposure. Combination ivTXA and tTXA has shown excellent results in total joint arthroplasty. The objective of this study is to determine the additive benefit and risks of co-administration of the two in spinal deformity surgery. This population of spinal patients was chosen because the estimated blood loss is high and the potential clinical benefit of the intervention is large. Patients will be enrolled if they are undergoing surgery > 5 levels with extension to the pelvis. The investigators have previously utilized topical TXA for these cases by applying operative sponges soaked with solution into the wound during routine x-ray check following instrumentation, with anecdotally good effect. However, this practice has not been prospectively studied. In this prospective, randomized, blinded, placebo controlled study, a similar combined effect of ivTXA and tTXA on decreasing perioperative blood loss as seen in total joint arthroplasty, with a similar safety profile is expected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Scheduled to undergo posterior long segment ( ≥ 5 levels) posterior spinal fusion for adult scoliosis or degenerative joint diseae
* + fusion to pelvis

Exclusion Criteria:

* Surgical factors:

  * Anterior Approach
  * Presence or history of dural tear without repair as evidenced by pseudomeningocele on MRI imaging or by intraoperative exploration
  * Patients donating autologous blood preoperatively

Patient factors:

* Diagnosis of renal (Cr>1.5 or CrCl <30ml/min) or hepatic insufficiency (AST, ALT 2x upper limit of normal)
* Diagnosis of seizure disorder or prior seizure
* History of thromboembolic events (CVA, TIA, DVT, PE) if within 1 year of surgery
* Hypercoagulability (e.g. antiphospholipid syndrome)
* History of coronary artery disease (stent, MI, +stress test) within 1 year of surgery
* Atrial fibrillation
* Concurrent anticoagulation therapy that cannot be discontinued within 3 days before surgery (Coumadin, plavix, LVX)
* Concurrent anticoagulation with ASA 325 that cannot be discontinued 10 days before surgery
* Bleeding disorder or abnormal preoperative coagulation profile (as identified by a preoperative platelet count of <100,000/mm3, an international normalized ratio of >1.4, or a prolonged partial thromboplastin time >1.4 times normal)
* Preexisting anemia <10 g/dL
* Color blindness or disturbance of color vision
* Leukemia or active cancer
* Religious restrictions on blood transfusion
* Pregnancy or women who are lactating/breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative Drain output | 48 hours
  Drain Output

SECONDARY OUTCOMES:
Perioperative blood transfusion | Up to 30 days postoperatively
  Number of units of blood transfused perioperatively, including cell saver administration
Perioperative blood drop | Up to 72 hours postoperatively
  CBC with hct/hg tracked postoperatively
Perioperative adverse events | Up to 30 days postoperatively
  Minor and major adverse events occuring during hospitalization or after discharge
Length of stay | Up to 30 days postoperatively
  # of days from surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Han Jo Kim, MD, Principal Investigator — Department of Spine Surgery
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No